CLINICAL TRIAL: NCT06222658
Title: The Role of Pharmaco-mechanical Thrombectomy in Management of Acute Lower Extremity Arterial Ischemia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Mohammed Rashed, dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PMT in acute limb ischemia
Record Dates: First submitted 2023-09-26; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Acute Limb Ischemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient assigned to pharmacomechanichal thrombectomy (Experimental)
  Interventions: Device: pharmaco-mechanichal thrombectomy

INTERVENTIONS:
Device: pharmaco-mechanichal thrombectomy — pharmaco-mechanichal thrombectomy in acute limb ischemia
  Other Names: Angiojet thrombectomy catheter

SUMMARY:
The goal of our protocol is to re-establish patency in ALLI, by combining both balloon maceration of a thrombus and angiojet PMT thus decreasing complications associated with prolonged periods of thrombolytic exposure while avoid open surgical risk .

DETAILED DESCRIPTION:
Acute lower extremity arterial ischemia (ALLI) is a common emergency in vascular surgery that has a high risk of limb amputation and mortality .It is caused by the blockage of an arterial flow to an extremity, which can be either thrombotic or embolic . Timely diagnosis and proper treatment for ALI are critical as to save limb viability .

Treatment options include surgical embolectomy, catheter-directed thrombolysis (CDT) , as well as pharmacochemical thrombectomy , Each of those approaches has its own disadvantages.

Fogarty manoeuvre embolectomy although flexible technique that can be used in a variety of situation, it is an open surgical procedure, carries the risk of complications such as bleeding and wound healing disorders. Additionally, it may impose a risk of arterial wall injury in the presence of underlying arterial lesions.

While CDT avoids common surgical complication its advantages include high risk of thrombo-lytic bleeding, residual thrombosis and long operation time and hospital stay.

As to address those limitations previous research has shown that using PMT as a first-line treatment for ALI provides rapid reperfusion to the extremity, reduces procedure time, and has an low risk profile .

The AngioJet Thrombectomy System (Boston Scientific Corporation, Marlborough, MA, USA) is a rheolytic PMT device that utilizes pressurized saline jets to generate a localized low-pressure zone (Bernoulli principle that results in fragmentation of the thrombus at the distal tip of the catheter.

The saline jets also provide the driving force through which the macerated thrombus particles are removed from the lesion site through the catheter. Several studies have demonstrated the effectiveness of the AngioJet system .

The goal of our protocol is to re-establish patency in ALLI, by combining both balloon maceration of a thrombus and angiojet PMT thus decreasing complications associated with prolonged periods of thrombolytic exposure while avoid open surgical risk .

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Symptom onset within 14 days for acute limb ischemia or within 30 days for subacute limb ischemia due to embolic or thrombotic occlusion of a native arteries, bypass graft, or arterial stent.

Rutherford category I, IIa or IIb

Exclusion Criteria:

* ALLI secondary to dissections, vasculitis, and/or target vessel trauma
* Pregnancy or positive pregnancy test
* Rutherford category III Irreversible (neglected) limb ischemia
* patients allergic to contrast agent,
* serum creatine>300 mmol/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2025-09-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Procedure success | immediately after angiography
  completion of the endovascular procedure without the need for further intervention for revascularization and an absence of substantial or complete occlusion in any vessel at final angiography
Amputation-free survival | 1 year
  freedom from amputation to the treated limb or mortality at follow-up at 30 days, 6 months and 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Asyut University Hospital, Asyut, Egypt

REFERENCES:
- [Background] Ascher E, Kibrik P, Rizvi SA, Alsheekh A, Marks N, Hingorani A. Fast-track thrombolysis protocol for acute limb ischemia. J Vasc Surg. 2021 Mar;73(3):950-959. doi: 10.1016/j.jvs.2020.03.061. Epub 2020 May 11. PMID 32437952
- [Background] Leung DA, Blitz LR, Nelson T, Amin A, Soukas PA, Nanjundappa A, Garcia MJ, Lookstein R, Simoni EJ. Rheolytic Pharmacomechanical Thrombectomy for the Management of Acute Limb Ischemia: Results From the PEARL Registry. J Endovasc Ther. 2015 Aug;22(4):546-57. doi: 10.1177/1526602815592849. Epub 2015 Jun 24. PMID 26109628
- See also: Rheolytic Pharmacomechanical Thrombectomy for the Management of Acute Limb Ischemia: Results From the PEARL Registry — https://pubmed.ncbi.nlm.nih.gov/26109628/
- See also: Fast-track thrombolysis protocol for acute limb ischemia — https://pubmed.ncbi.nlm.nih.gov/32437952/